CLINICAL TRIAL: NCT00465049
Title: Primary vs. Secondary Closure of Cutaneous Abscesses After I&D: A RCT
Brief Title: Comparison of Suturing and Packing of Drained Abscesses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, RESEARCH DIRECTOR, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORIHS 2007-5819
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Cutanoeus Abscesses
Keywords: abscess, primary closure, secondary closure
MeSH Terms: conditions — Abscess

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- primary closure (Experimental): suture after I&D
  Interventions: Other: PRIMARY CLOSRE
- SECONDARY CLOSURE (Placebo Comparator): LEAVE TO HEAL BY SECONDARY INTENTIN AFTER I&D
  Interventions: Other: SECONDARY CLOSURE; Other: SPONTANEOUS HALING

INTERVENTIONS:
Other: PRIMARY CLOSRE — SUTURE
  Arms: primary closure
Other: SECONDARY CLOSURE — ALLOW TO HEAL SPONTANEOUSLY
  Arms: SECONDARY CLOSURE
Other: SPONTANEOUS HALING — SECONDARY HEALING AFTER I&D
  Arms: SECONDARY CLOSURE

SUMMARY:
The standard treatment for skin abscesses in drainage followed by packing to prevent premature closure and reaccumulation of pus. Studies from the 1950s and later conducted outside of the US suggest that when drained abscesses are drained and sutured closed they actually heal faster without complications. The current study compares the time to healing and scar formation when drained abscesses are packed or sutured.

ELIGIBILITY:
Inclusion Criteria:

* Non complicated abscesses

Exclusion Criteria:

* Fever,
* Immunocompromise,
* Cellulitis,
* Perianal and
* Pilonidal abscesses

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Days to healing. | 1 week

SECONDARY OUTCOMES:
Need for subsequent drainage, scar appearance. | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Adam J Singer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

REFERENCES:
- [Background] ELLIS M. Incision and primary suture of abscesses of the anal region. Proc R Soc Med. 1960 Aug;53(8):652-3. doi: 10.1177/003591576005300819. No abstract available. PMID 13726484
- [Background] Khanna YK, Khanna A, Singh SP, Laddha BL, Prasad P, Jhanji RN. Primary closure of gluteal injection abscess (a study of 100 cases). J Postgrad Med. 1984 Apr;30(2):105-10. No abstract available. PMID 6527292
- [Background] Ajao OG, Ladipo JK, al-Saigh AA, Malatani T. Primary closure of breast abscess compared with the conventional gauze packing and daily dressings. West Afr J Med. 1994 Jan-Mar;13(1):28-30. PMID 8080827
- [Background] Stewart MP, Laing MR, Krukowski ZH. Treatment of acute abscesses by incision, curettage and primary suture without antibiotics: a controlled clinical trial. Br J Surg. 1985 Jan;72(1):66-7. doi: 10.1002/bjs.1800720125. PMID 3881155
- [Background] Edino ST, Ihezue CH, Obekpa PO. Outcome of primary closure of incised acute soft-tissue abscesses. Niger Postgrad Med J. 2001 Mar;8(1):32-6. PMID 11487781
- [Background] Abraham N, Doudle M, Carson P. Open versus closed surgical treatment of abscesses: a controlled clinical trial. Aust N Z J Surg. 1997 Apr;67(4):173-6. doi: 10.1111/j.1445-2197.1997.tb01934.x. PMID 9137156
- [Derived] Singer AJ, Taira BR, Chale S, Bhat R, Kennedy D, Schmitz G. Primary versus secondary closure of cutaneous abscesses in the emergency department: a randomized controlled trial. Acad Emerg Med. 2013 Jan;20(1):27-32. doi: 10.1111/acem.12053. PMID 23570475